CLINICAL TRIAL: NCT00096928
Title: Raptiva Epidemiologic Study of Psoriasis Outcomes and Safety Events in Patients With Chronic Moderate to Severe Plaque Psoriasis (RESPONSE)
Brief Title: A Study to Evaluate Psoriasis Outcomes and Safety Events in Patients With Chronic Moderate to Severe Plaque Psoriasis (RESPONSE)
Acronym: RESPONSE
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Disclosures Group, Genentech, Inc.
Other Study IDs: ACD3101g
Record Dates: First submitted 2004-11-17; First posted 2004-11-18 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2011-03

CONDITIONS: Psoriasis
Keywords: Plaque Psoriasis; RESPONSE; Raptiva; efalizumab
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This was a multicenter, prospective, 5-year surveillance study of approximately 5000 Raptiva-treated patients and approximately 500 non-Raptiva treated patients (formerly 2500 comparison patients who were treated with a biologic therapy other than Raptiva) with chronic moderate to severe plaque psoriasis who were candidates for treatment with Raptiva.

ELIGIBILITY:
Inclusion Criteria:

* Have ever had a physician's diagnosis of chronic moderate to severe plaque psoriasis and be a candidate for treatment with Raptiva
* Are being treated with or initiating Raptiva therapy at the time of enrollment
* Be able to provide written informed consent
* Be willing and able to fully to participate for the duration of patient follow-up (5 years)

Exclusion Criterion:

* Have previously received at least one dose of Raptiva and are not currently using or restarting treatment with Raptiva at the time of enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: managed care organizations, community or physician practices, and academic centers in the United States
Sampling Method: Probability Sample
Enrollment: 1846 (Actual)
Dates: Start 2005-03; Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivor Caro, M.D., Study Director — Genentech, Inc.
Locations (182):
- United States (182):
  - Total Skin and Beauty Dermatology Center, Birmingham, Alabama
  - Deep South Dermatology, Daphne, Alabama
  - The Dermatology Center, Gadsden, Alabama
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - Ruth A. Yates, MD, Huntsville, Alabama
  - SunValley Arthritis Center Ltd, Glendale, Arizona
  - Alliance Dermatology and MOHS, Phoenix, Arizona
  - BGPDS Dermatology, Little Rock, Arkansas
  - Hull Dermatology, PA, Rogers, Arkansas
  - Bakersfield Dermatology and Skin Cancer Medical Grp, Bakersfield, California
  - T. Joseph Raoof, MD, Inc., Encino, California
  - Minarets Medical Group, Fresno, California
  - Associates In Research, Inc., Fresno, California
  - Delta Dermatology Medical Group, Inglewood, California
  - Fairmont Dermatology Medical Associates, Inc, Lodi, California
  - Dermatology Associates, Los Angeles, California
  - Elizabeth A. Abel, MD, Mountain View, California
  - Dermatology Medical Group of Oxnard, Oxnard, California
  - Kent Carson, MD, San Jose, California
  - East Bay Psoriasis Treatment Center, San Ramon, California
  - Clinical Research Specialists, Inc., Santa Monica, California
  - Healthcare Partners Medical Group, Torrance, California
  - Skin Physicians and Surgeons Medical Group, Inc., Upland, California
  - Centennial Cosmetic Surgery and Dermatology, Centennial, Colorado
  - Colorado Medical Research Center, Inc., Denver, Colorado
  - Meridian Skin Cancer Center, Englewood, Colorado
  - Northern Colorado Allergy and Asthma Clinic, Greeley, Colorado
  - Dermatology Associates Of Western Connecticut, Danbury, Connecticut
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Aventura Medical Research Inc, Aventura, Florida
  - Stephen N Horwitz, MD, PA, Aventura, Florida
  - Brent M Schillinger, MD, PA, Boca Raton, Florida
  - The Dermatology and Aesthetic Center, Boca Raton, Florida
  - David Hecker, MD, Boca Raton, Florida
  - Dermatology Associates and Research, Coral Gables, Florida
  - North Florida Dermatology Associates, PA, Jacksonville, Florida
  - Coastal Dermatology, Jacksonville, Florida
  - Genesis Dermatology, Jupiter, Florida
  - University of Miami Dept. of Dermatology and Cutaneous Surgery, Miami, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - Central Florida Dermatology Associates, Inc., Orlando, Florida
  - Dermatology Consultants of Broward, Pembroke Pines, Florida
  - Dermatology Research by Dr. Gary L. Heller, Pinellas Park, Florida
  - Clinical Research of Tampa Bay, Inc., Spring Hill, Florida
  - Atlanta Dermatology, Vein, and Research Center, LLC, Alpharetta, Georgia
  - Emory University, Atlanta, Georgia
  - Dermatology Specialists of West Georgia, Carrollton, Georgia
  - East Metro Dermatology, Conyers, Georgia
  - Dermatologic Surgery Specialists, Inc., Macon, Georgia
  - Northwest Georgia Dermatology, Rome, Georgia
  - Gwinnett Clinical Research Center Inc., Snellville, Georgia
  - Toccoa Clinic Medical Associates, Toccoa, Georgia
  - Queens Medical Center, Honolulu, Hawaii
  - Alan Olmstead, MD, Twin Falls, Idaho
  - Fox Valley Dermatology LTD, Aurora, Illinois
  - Christie Clinic, Champaign, Illinois
  - Northwestern University, Chicago, Illinois
  - Danilo V. Del Campo, Chicago, Illinois
  - Advanced Dermatology, Lincolnshire, Illinois
  - Skin Care Center Of Southern Illinois, Mount Vernon, Illinois
  - Schaumburg Dermatology, Schaumburg, Illinois
  - Dermatology Center of Northwest Indiana, Crown Point, Indiana
  - Three Rivers Dermatology, Fort Wayne, Indiana
  - Dermatology Associates, PC, Indianapolis, Indiana
  - Investigators Research Group, Indianapolis, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The Dermatology Center PSC, New Albany, Indiana
  - The Dermatology Center of Indiana, Plainfield, Indiana
  - Randall Dermatology, PC, West Lafayette, Indiana
  - University of Iowa Health Care, Iowa City, Iowa
  - Kansas City Dermatology, PA, Overland Park, Kansas
  - Kansas Medical Clinic, Topeka, Kansas
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - Derm Research, PLLC, Louisville, Kentucky
  - Louisiana Dermatology Associates, Baton Rouge, Louisiana
  - Dermatology and Advanced Aesthetics, Lake Charles, Louisiana
  - Highland Clinic, APMC, Shreveport, Louisiana
  - Washington Dermatology Center, Bethesda, Maryland
  - Callender Skin and Laser Center, Mitchellville, Maryland
  - Brigham and Womens' Hospital, Boston, Massachusetts
  - Skin Care Physicians of Chestnut Hill, Chestnut Hill, Massachusetts
  - Dermatology Associates, Norwood, Massachusetts
  - Worcester Dermatology, Worcester, Massachusetts
  - David Fivenson, MD Dermatology, PLLC, Ann Arbor, Michigan
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Psoriasis and Eczema Treatment Center of Western Michigan PLLC, Grand Rapids, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - M. Siegel, MD PC, Waterford, Michigan
  - Lloyd J. Cleaver, DO, LLC, Kirksville, Missouri
  - Saint Louis University, St Louis, Missouri
  - Central Dermatology, PC, St Louis, Missouri
  - Jacquelyn B. Garrett, St Louis, Missouri
  - Karen E Forsman, MD Dermatology LLC, St Louis, Missouri
  - South Lincoln Dermatology, Lincoln, Nebraska
  - Woodson Dermatology, Las Vegas, Nevada
  - Nevada Center For Dermatology, Ltd, Reno, Nevada
  - Skin Cancer and Dermatology Institute, Reno, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Nashua Dermatology Associates, Nashua, New Hampshire
  - Nashua Dermatology, Nashua, New Hampshire
  - Belleville Dermatology Ctr, PA, Belleville, New Jersey
  - Windsor Dermatology, East Windsor, New Jersey
  - Hudson Dermatology and Skin Cancer Center, Hoboken, New Jersey
  - Karen S. Harkaway, MD, LLC, Riverside Park, New Jersey
  - Associates In Dermatology Research, Rutherford, New Jersey
  - Linda Susan Marcus, MD, FAAD, Wyckoff, New Jersey
  - The Dermatology Center, Bayside, New York
  - Jeffrey Schachne, MD, Jefferson Valley, New York
  - Atlantic Dermatologic Associates, LLP, Lynbrook, New York
  - DiGiovanna Family Care Center, North Massapequa, New York
  - South Nassau Dermatology, P.C., Oceanside, New York
  - Helendale Dermatology and Medical Spa, Rochester, New York
  - Skin Search and Dermatology Associates of Rochester, Rochester, New York
  - The Center for Dermatology at Lifetime Health, Rochester, New York
  - Thomas O. McMeekin MD, PC, Rochester, New York
  - Dermatology Associates, Staten Island, New York
  - DermResearchCenter of New York, Inc, Stony Brook, New York
  - Arthritis Health Associates, Syracuse, New York
  - Buffalo Medical Group, PC, Williamsville, New York
  - Mid-Charlotte Dermatology and Research PLLC, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Dermatology and Skin Cancer Center, Raleigh, North Carolina
  - Andrus and Associates Dermatology, P.A., Raleigh, North Carolina
  - Atlantic Dermatology Associates PA, Wilmington, North Carolina
  - Wilmington Health Associates, Wilmington, North Carolina
  - Curtis W. Hawkins, MD, Akron, Ohio
  - DataPharm, Inc., Canfield, Ohio
  - University Dermatology Consultants, Inc., Cincinnati, Ohio
  - University Hospitals Cleveland, Cleveland, Ohio
  - The Cleveland Clinical Foundation, Cleveland, Ohio
  - Wright State University, Dayton, Ohio
  - Hudson Dermatology, Hudson, Ohio
  - Wells Institute for Health Awareness, Kettering, Ohio
  - Smith Clinic, Marion, Ohio
  - Jan Fu, MD and PhD, Mason, Ohio
  - Judith Andreano MD, Inc., Strongsville, Ohio
  - DataPharm, Inc, Warren, Ohio
  - Sooner Palmer Circle, Norman, Oklahoma
  - Northwest Cutaneous Research Specialists, Portland, Oregon
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Jan K. Brydon, MD, Erie, Pennsylvania
  - Atlantic Skin and Cosmetic Surgery Group, PC, Malvern, Pennsylvania
  - East Penn. Dermatology, North Wales, Pennsylvania
  - Dermatology Associates Of Plymouth Meeting, Plymouth Meeting, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Dermatology Associates of the Low Country, Beaufort, South Carolina
  - Dr. Marta Hampton, Charleston, South Carolina
  - Dermatology and Laser Center of Charleston, PA, Charleston, South Carolina
  - Advanced Dermatology and Laser Center, Greenville, South Carolina
  - Germain Dermatology Associates, Mt. Pleasant, South Carolina
  - The Hillcrest Dermatology Center, Orangeburg, South Carolina
  - Southeastern Research Associates, Inc., Taylors, South Carolina
  - Dakota Dermatology, LTD, Sioux Falls, South Dakota
  - James E. Turner, MD, PhD, PC, Bartlett, Tennessee
  - Advanced Skin and Laser Center, Brentwood, Tennessee
  - Rivergate Dermatology, Goodlettsville, Tennessee
  - Dermatology Associates of Kingsport, PC, Kingsport, Tennessee
  - Dermatology Associates Of Knoxville, Knoxville, Tennessee
  - The Skin Wellness Center, P.C., Knoxville, Tennessee
  - Murfreesboro Dermatology Clinic, Murfreesboro, Tennessee
  - Dermatology Research Associates Inc., Nashville, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Familicare Clinical Research, Colleyville, Texas
  - Baylor Research Institute, Dallas, Texas
  - West Houston Dermatology, PA, Houston, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Dermatology Associates of San Antonio, San Antonio, Texas
  - Rocky Mountain Dermatology, Logan, Utah
  - Fletcher Allen Health Care, Burlington, Vermont
  - Education and Research Foundation, Lynchburg, Virginia
  - Virginia Clinical Research, Norfolk, Virginia
  - Skin and Laser Surgery Center PC, Tysons Corner, Virginia
  - Virginia Beach Dermatology Associates, Virginia Beach, Virginia
  - Dermatology Associates, Inc., Winchester, Virginia
  - Dermatology and Laser Center NW, Bellingham, Washington
  - Eastern Washington Dermatology, Dayton, Washington
  - Dermatology Associates, PLLC, Seattle, Washington
  - Spokane Dermatology Clinic, Spokane, Washington
  - Northwest Dermatology, Spokane, Washington
  - Great Lakes Dermatology- Racine, Racine, Wisconsin
  - Aylesworth Dermatology, SC, Rhinelander, Wisconsin